CLINICAL TRIAL: NCT04955951
Title: Ultrasonographic Response to Polarized Light Therapy in the Treatment of Atopic Dermatitis
Status: Terminated | Type: Observational
Why Stopped: forgotten
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mahmoud H Mohamed, PhD, LECTURER, Ahram Canadian University
Other Study IDs: AhramCUE
Record Dates: First submitted 2021-06-16; First posted 2021-07-09 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2021-10

CONDITIONS: Chronic Atopic Dermatitis
MeSH Terms: interventions — Microscopy, Polarization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- polarized light group: group A (20 patients) will receive Polarized light therapy
  Interventions: Device: polarized light
- topical corticosteroid group: group B (20 patients) will receive topical corticosteroid therapy
  Interventions: Drug: Topical corticosteroid ointment

INTERVENTIONS:
Device: polarized light — A Bioptron light therapy phototherapeutic device (Bioptron AG, Wollerau, Switzerland) with 5 cm treatment diameter (BIOPTRON MedAll®, 480-3400 nm, polarization level of 95%, power density 40 mW/cm2, energy density 2,4 J/cm2 per minute
  Groups: polarized light group
Drug: Topical corticosteroid ointment — corticosteroid 1 %.
  Groups: topical corticosteroid group

SUMMARY:
Non-atopic dermatitis (NAD) or eczema is a common inflammatory condition; potentially debilitating that can compromise quality of life. It is usually seen in childhood, but can onset within or persist into adulthood.

DETAILED DESCRIPTION:
Polarized ultraviolet-free polychromatic light is used as therapeutic option for the treatment of wound healing and dermatological conditions.

40 male patients who had atopic dermatitis in the chronic stage, they were complaining from itching, inflammation and skin thickness in the arm, wrist, hand and leg will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* The patients' ages will ranged from 20 to 30 years.
* The subjects will be males.
* The duration of disease less than 1 year.

Exclusion Criteria:

* patients who had skin malignancy in the area to be treated.
* The patients who had history of diabetes, circulatory or sensory disorders.
* Patients with acute infection in the area treated.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20-30
Study Population: The Patient will be referred to physical therapy outpatient clinic, faculty of physical therapy, Ahram Canadian University from dermatology out-clinics in Sheikh Zayed Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Ultrasonography | 1-2 months
  Ultrasound imaging system used to measure the thickness of the skin at the site of scale for both groups

SECONDARY OUTCOMES:
SCORAD Score | 1-2 months
  The SCORAD (Index) is the best validated scoring system in atopic dermatitis, To measure the extent of AD, the rule of nines is applied on a front/back drawing of the patient's inflammatory lesions. The extent can be graded from 0 to 100. The intensity part of the SCORAD consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness. Each item can be graded on a scale from 0 to 3. The subjective items include daily pruritus and sleeplessness. The SCORAD Index formula is: A/5 + 7B/2 + C. In this formula A is defined as the extent (0-100), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The maximal score of the SCORAD Index is 103. The objective SCORAD consist of the extent and the intensity items; the formula is A/5 + 7B/2. The maximal objective SCORAD score is 83 (with 10 additional points for severe disfiguring eczema of the face and hands).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Canadian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
ultrasonographic skin thickness results will be shared